CLINICAL TRIAL: NCT00839917
Title: A Multicenter, Randomized, Open-Label Study to Compare the Immunogenicity, Safety, and Tolerability of Measles, Mumps, Rubella, and Varicella of Combination Vaccine ProQuad With Concomitant Administration of M-M-R II and VARIVAX in Healthy Korean Children
Brief Title: A Study of ProQuad™ in Healthy Children in Korea (V221-023)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early because of insufficient enrollment before expiration date of the investigational vaccine lot
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-023; 2009_538
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Measles; Mumps; Rubella; Varicella
Keywords: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine; Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProQuad™ (Experimental)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live (ProQuad™)
- M-M-R™ II and Varivax™ (Active Comparator)
  Interventions: Biological: M-M-R™ II and Varivax™

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live (ProQuad™) — Single administration of 0.5 mL subcutaneous injection
  Other Names: V221
  Arms: ProQuad™
Biological: M-M-R™ II and Varivax™ — Single administration of 0.5 mL subcutaneous injection
  Arms: M-M-R™ II and Varivax™

SUMMARY:
This study will compare ProQuad™ and concomitant administration of M-M-R™ II and Varivax™ with respect to immunogenicity, safety and tolerability. The primary hypothesis to be tested is that the antibody response rates to measles, mumps, rubella, and varicella 6 weeks after vaccination with ProQuad™ will be non-inferior to the antibody response rates after vaccination with concomitant M-M-R™ II and Varivax™.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject has a negative clinical history for measles, mumps, rubella, varicella and zoster

Exclusion Criteria:

* Subject has previously received measles, mumps, rubella and/or varicella vaccine, either alone or in any combination
* Subject has any congenital or acquired immune deficiency, neoplastic disease or depressed immunity
* Subject has a history of seizure disorder
* Subject had exposure to measles, mumps, rubella, varicella and/or zoster in the last 4 weeks
* Subject has received an inactivated vaccine within the past 14 days
* Subject has received a live vaccine within the past 30 days
* Subject has received immune globulin within the past 5 months
* Subject has a recent history of fever (within the last 72 hours)

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to enroll 360 participants; however the study was terminated early because it was not possible to complete enrollment before expiration of the investigational vaccine lot
Groups:
- ProQuad™; M-M-R™ II and Varivax™: Single subcutaneous 0.5 mL vaccination
Period: Overall Study
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Started | 13 | 17
Completed | 12 (Study completers were randomized participants who received study vaccination and had follow-up data) | 16 (Study completers were randomized participants who received study vaccination and had follow-up data)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did not receive vaccine | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™ | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Customized [Number; unit: participants]
  12 to 15 months | 13 | 17 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Measles Antibody Levels ≥255 mIU/mL
Description: Antibody response to measles at 6 weeks after vaccination for participants initially seronegative (<255 mIU/mL) to measles at baseline
Time Frame: 6 weeks postvaccination
Population: Analysis was performed on the per-protocol population, defined as all participants who had both pre- and post-vaccination blood samples, were seronegative at baseline, and followed all protocol procedures. Too few participants were enrolled in the study to perform non-inferiority analysis for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
percentage of participants | 100.0 [74.1 to 100.0] | 87.5 [52.9 to 99.4]

2. Primary Outcome: Percentage of Participants With Mumps Antibody Levels ≥10 Mumps Antibody Units/mL
Description: Antibody response to mumps at 6 weeks after vaccination for participants initially seronegative (<10 units/mL) to mumps at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
percentage of participants | 100.0 [74.1 to 100.0] | 100.0 [68.8 to 100.0]

3. Primary Outcome: Percentage of Participants With Rubella Antibody Levels ≥10 IU/mL
Description: Antibody response to rubella at 6 weeks after vaccination for participants initially seronegative (<10 IU/mL) to rubella at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
percentage of participants | 100.0 [74.1 to 100.0] | 100.0 [68.8 to 100.0]

4. Primary Outcome: Percentage of Participants With Varicella-zoster Virus (VZV) Antibody Levels ≥5 Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Units/mL
Description: Antibody response to VZV at 6 weeks after vaccination for participants initially seronegative (<5 gpELISA units/mL) to VZV at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
percentage of participants | 90.0 [60.6 to 99.5] | 100.0 [68.8 to 100.0]

5. Secondary Outcome: Geometric Mean Titer of Measles Antibodies
Description: Mean measles antibody response at 6 weeks after vaccination for participants initially seronegative (<255 mIU/mL) to measles at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: mIU/mL
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
mIU/mL | 5270.7 [3952.0 to 7029.3] | 3516.2 [1188.8 to 10396.5]

6. Secondary Outcome: Geometric Mean Titer of Mumps Antibodies
Description: Mean mumps antibody response at 6 weeks after vaccination for participants initially seronegative (<10 Units/mL) to mumps at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: Units/mL
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
Units/mL | 159.2 [93.1 to 271.8] | 104.4 [59.2 to 183.5]

7. Secondary Outcome: Geometric Mean Titer of Rubella Antibodies
Description: Mean rubella antibody response at 6 weeks postvaccination for participants initially seronegative (<10 IU/mL) to rubella at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: IU/mL
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
IU/mL | 105.8 [69.6 to 160.5] | 147.1 [105.6 to 204.9]

8. Secondary Outcome: Geometric Mean Titer of VZV (gpELISA) Antibodies
Description: Mean VZV antibody response at 6 weeks after vaccination for participants initially seronegative (<5 gpELISA Units/mL) to VZV at baseline
Time Frame: 6 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: gpELISA units/mL
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 10 | 8
gpELISA units/mL | 10.4 [6.9 to 15.5] | 11.9 [7.6 to 18.4]

9. Other Pre Specified Outcome: Percentage of Participants With Measles-like Rash
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 0.0 | 12.5

10. Other Pre Specified Outcome: Percentage of Participants With Varicella-like Rash
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 0.0 | 0.0

11. Other Pre Specified Outcome: Percentage of Participants With Rubella-like Rash
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 0.0 | 0.0

12. Other Pre Specified Outcome: Percentage of Participants With Zoster-like Rash
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 0.0 | 0.0

13. Other Pre Specified Outcome: Percentage of Participants With Any Systemic Adverse Experience
Description: An adverse experience is defined as any unfavorable and unintended change in the
  structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse experience. A systemic adverse experience is any adverse experience other than injection-site adverse experiences.
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 53.9 | 56.3

14. Other Pre Specified Outcome: Percentage of Participants With Injection-site Adverse Experiences
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse experience. An injection-site adverse experience is an adverse experience that occurs at the injection site only.
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 15.4 | 0.0

15. Other Pre Specified Outcome: Percentage of Participants With Injection-site Adverse Experiences
Description: as for outcome 14
Time Frame: Through 5 days postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 7.7 | 0.0

16. Other Pre Specified Outcome: Percentage of Participants With Fever (≥101.0°F [38.3°C] Axillary or ≥103.0°F [39.4°C] Rectal)
Time Frame: Through 6 weeks postvaccination
Population: The safety population included all participants who received study vaccination
Measure: Number; unit: percentage of participants
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Number analyzed (Participants) | 13 | 16
percentage of participants | 7.7 | 12.5

ADVERSE EVENTS:
Time Frame: Through 28 days postvaccination
Description: The safety population included all participants who received study vaccination
Arm/Group | ProQuad™ | M-M-R™ II and Varivax™
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/16
Other Adverse Events (participants affected / at risk) | 8/13 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProQuad™ (N=13) | M-M-R™ II and Varivax™ (N=16)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProQuad™ (N=13) | M-M-R™ II and Varivax™ (N=16)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (4)
Swelling (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (3) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Formal testing of the study hypotheses was not possible because of low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.